CLINICAL TRIAL: NCT05010772
Title: Oral Decitabine-Based Maintenance Therapy in Patients With AML in Remission
Brief Title: Decitabine Alone or in Combination With Venetoclax, Gilteritinib, Enasidenib, or Ivosidenib as Maintenance Therapy for the Treatment of Acute Myeloid Leukemia in Remission
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021-0237; NCI-2021-08496 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2021-0237 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2021-08-11; First posted 2021-08-18 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — decitabine and cedazuridine drug combination; enasidenib; gilteritinib; ivosidenib; venetoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (5):
- Arm A (decitabine and cedazuridine) (Experimental): Patients receive decitabine and cedazuridine PO QD on days 1-3. Treatments repeat every 28 days for up to 4 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Decitabine and Cedazuridine
- Arm B (decitabine and cedazuridine, venetoclax) (Experimental): Patients receive decitabine and cedazuridine PO QD on days 1-3 and venetoclax PO QD on days 1-5. Treatments repeat every 4 weeks for up to 24 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Decitabine and Cedazuridine; Drug: Venetoclax
- Arm C (decitabine and cedazuridine, gilteritinib) (Experimental): Patients receive decitabine and cedazuridine PO QD on days 1-3 and gilteritinib PO QD on days 1-28. Treatments repeat every 4 weeks for up to 24 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Decitabine and Cedazuridine; Drug: Gilteritinib
- Arm D (decitabine and cedazuridine, enasidenib) (Experimental): Patients receive decitabine and cedazuridine PO QD on days 1-3 and enasidenib PO QD on days 1-28. Treatments repeat every 4 weeks for up to 24 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Decitabine and Cedazuridine; Drug: Enasidenib
- Arm E (decitabine and cedazuridine, ivosidenib) (Experimental): Patients receive decitabine and cedazuridine PO QD on days 1-3 and ivosidenib PO QD on days 1-28. Treatments repeat every 4 weeks for up to 24 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Decitabine and Cedazuridine; Drug: Ivosidenib

INTERVENTIONS:
Drug: Decitabine and Cedazuridine — Given PO
  Other Names: ASTX727; C-DEC; CDA Inhibitor E7727/Decitabine Combination Agent ASTX727; Cedazuridine/Decitabine Combination Agent ASTX727; Cedazuridine/Decitabine Tablet; DEC-C; Inqovi
Drug: Enasidenib — Given PO
  Other Names: AG-221; CC-90007 Free Base
  Arms: Arm D (decitabine and cedazuridine, enasidenib)
Drug: Gilteritinib — Given PO
  Other Names: ASP-2215; ASP2215
  Arms: Arm C (decitabine and cedazuridine, gilteritinib)
Drug: Ivosidenib — Given PO
  Other Names: AG-120; Tibsovo
  Arms: Arm E (decitabine and cedazuridine, ivosidenib)
Drug: Venetoclax — Given PO
  Other Names: ABT-0199; ABT-199; ABT199; GDC-0199; RG7601; Venclexta; Venclyxto
  Arms: Arm B (decitabine and cedazuridine, venetoclax)

SUMMARY:
This phase Ib trial is to find out the side effects and possible benefits of decitabine alone or given together with venetoclax, gilteritinib, enasidenib, or ivosidenib in treating patients with acute myeloid leukemia that is under control (remission). Chemotherapy drugs, such as decitabine, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Venetoclax may stop the growth of cancer cells by blocking a protein called Bcl-2 needed for cell growth. Gilteritinib, enasidenib, and ivosidenib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Giving decitabine alone or together with venetoclax, gilteritinib, enasidenib, or ivosidenib may help to control the disease.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To assess safety of patients with acute myeloid leukemia (AML) treated with decitabine and cedazuridine (oral decitabine)-based combinations as maintenance therapy after achieving remission.

SECONDARY OBJECTIVES:

I. To assess relapse-frees survival (RFS) of patients with AML treated with oral decitabine-based combinations as maintenance therapy.

II. To assess overall survival (OS) of patients with AML treated with oral decitabine-based combinations as maintenance therapy.

III. To assess event-free survival (EFS) of patients with AML treated with oral decitabine-based combinations as maintenance therapy.

IV. To assess the duration of remission (CRd) of patients with AML treated oral decitabine-based combinations as maintenance therapy.

V. To assess the effects of oral decitabine-based combinations on dynamics of minimal residual disease and their relationship to outcomes.

EXPLORATORY OBJECTIVE:

I. To evaluate RFS in (1) intensive induction cohort and (2) lower intensity induction cohort.

OUTLINE: Patients are assigned to 1 of 5 arms.

ARM A: Patients receive decitabine and cedazuridine orally (PO) once daily (QD) on days 1-3. Treatments repeat every 28 days for up to 4 weeks in the absence of disease progression or unacceptable toxicity.

ARM B: Patients receive decitabine and cedazuridine PO QD on days 1-3 and venetoclax PO QD on days 1-5. Treatments repeat every 4 weeks for up to 24 cycles in the absence of disease progression or unacceptable toxicity.

ARM C: Patients receive decitabine and cedazuridine PO QD on days 1-3 and gilteritinib PO QD on days 1-28. Treatments repeat every 4 weeks for up to 24 cycles in the absence of disease progression or unacceptable toxicity.

ARM D: Patients receive decitabine and cedazuridine PO QD on days 1-3 and enasidenib PO QD on days 1-28. Treatments repeat every 4 weeks for up to 24 cycles in the absence of disease progression or unacceptable toxicity.

ARM E: Patients receive decitabine and cedazuridine PO QD on days 1-3 and ivosidenib PO QD on days 1-28. Treatments repeat every 4 weeks for up to 24 cycles in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 6-12 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged >= 18 years AML who have achieved their FIRST complete response (CR) or complete response with incomplete bone marrow recovery (CRi) and are not immediately candidates for allogeneic stem cell transplant
* Patients who have received intensive therapy (defined as receiving standard or higher dose cytarabine-based therapy) to achieve remission (CR/CRi) should have received remission induction therapy and at least 1 consolidation cycle. These patients are eligible as long as they are not greater than 2 months from their last consolidation therapy and will be designated as COHORT 1 (intensive induction cohort)
* Patients who have received lower intensity therapy (defined as receiving low-dose cytarabine [LDAC] or hypomethylating agent [HMA]-based therapy) to achieve remission should have received at least 2 cycles of lower intensity therapy between the time they have achieved CR/CRi and enrollment on this protocol. They will be designated as COHORT 2 (lower intensity induction cohort)
* For either subgroup (lower or higher intensity), patients who have measurable residual disease may be enrolled on their respective cohort at any time without maximum 'time from consolidation' requirement
* Eastern Cooperative Oncology Group (ECOG) performance status of < or = 3
* Serum total bilirubin < or = to 1.5 x the upper limit of normal (ULN)
* Serum creatinine < or = to 2.5 x ULN
* Absolute neutrophil count (ANC) > 0.5 x k/uL
* Platelet count > or = 50 x k/uL
* For females of childbearing age, they may participate if they:

  * Have a negative serum or urine pregnancy test within 10 to 14 days of enrolling
  * Agree to either abstinence or 2 effective contraceptive methods (such as barrier methods or hormonal contraception) throughout the treatment period and up to 30 days after discontinuing treatment
* For male patients with a female partner of childbearing age, they may participate if they agree to either abstinence or 2 effective contraceptive methods throughout the treatment period and up to 30 days after discontinuing treatment
* Ability to understand and sign informed consent

Exclusion Criteria:

* Diagnosis of acute promyelocytic leukemia (APL), AML - M3 by French-American-British (FAB) classification based on morphology, immunophenotype, molecular, or cytogenetics studies
* Diagnosis of AML associated t(15;17) or APL variant. Patients with t(9;22) are also ineligible unless they are unable or unwilling to receive therapy with a tyrosine kinase inhibitor
* Uncontrolled intercurrent illness including, but not limited to active uncontrolled infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Patients with active CNS (central nervous system) disease
* Patients with documented hypersensitivity to any components of the study program
* Females who are pregnant or lactating or intending to become pregnant during the study
* Patients with history of extramedullary AML, except for CNS involvement that is currently controlled, will not be eligible for enrollment
* Patient should be removed from current trial if they wish to participate and get treatment on another trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Estimated)
Dates: Start 2021-10-25 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events | Up to 5 years
  Safety analyses in general will be descriptive and will be presented in tabular format with the appropriate summary statistics. Adverse events will be tabulated using frequency and percentage by severity and by relations to the treatments for each arm.

SECONDARY OUTCOMES:
Relapse-free survival (RFS) | From complete remission or complete remission with incomplete count recovery until date of first objective documentation of relapse or death, assessed up to 5 years
  The Kaplan-Meier method will be used to estimate RFS.
Overall survival (OS) | From date of treatment start until date of death due to any cause, assessed up to 5 years
  The Kaplan-Meier method will be used to estimate OS.
Event-free survival (EFS) | From treatment start until date of first documented event., assessed up to 5 years
  Event will be defined as: confirmed relapse, withdrawal from study due to adverse event, or death due to any cause. The Kaplan-Meier method will be used to estimate EFS.
Duration of remission | Up to 5 years
  The Kaplan-Meier method will be used to duration of remission.
Minimal residual disease | Up to 5 years
  The log rank test and Cox proportional hazards model will be used to evaluate the association between the time to event outcomes and status of residual disease.

OTHER OUTCOMES:
RFS (Intensive induction cohort) | Up to 5 years
  Kaplan-Meier method will be used to estimate RFS for intensive induction cohort.
RFS (Lower intensity induction cohort) | Up to 5 years
  Kaplan-Meier method will be used to estimate RFS for lower intensity induction cohort.

CONTACTS AND LOCATIONS:
Overall Officials: Tapan M Kadia, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org